CLINICAL TRIAL: NCT00002431
Title: A Multi-Center Trial to Evaluate the Safety and Effectiveness of Peridex Dosed Twice or Three Times Daily for Preventing or Delaying the Occurrence of Lesions Due to Oral Candidiasis in HIV-Positive Individuals
Brief Title: The Safety and Effectiveness of Peridex in Preventing or Delaying Fungal Infections of the Mouth in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 050A; CC-220
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-11

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; chlorhexidine gluconate; Acquired Immunodeficiency Syndrome; Anti-Infective Agents, Local; AIDS-Related Complex; Candidiasis, Oral
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — chlorhexidine gluconate

INTERVENTIONS:
Drug: Chlorhexidine gluconate

SUMMARY:
To evaluate the safety and effectiveness of Peridex (an oral rinse containing chlorhexidine gluconate) for preventing the occurrence of clinically-evident microbiologically-documented oral candidiasis in HIV-positive patients, who are at risk of the disease based on previous history of candidiasis.

ELIGIBILITY:
Inclusion Criteria

Prior Medication:

Allowed within 6 months of study entry:

* Treatment for oral candidiasis.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Either history of esophageal candidiasis or current mucocutaneous candidiasis (angular cheilitis).
* Allergies to chlorhexidine.
* Gross periodontal neglect or need for periodontal treatment within the past two weeks.

Concurrent Medication:

Excluded:

* Systemic or oral topical mucocutaneous antifungal therapy.
* Systemic or oral topical corticosteroids.
* Antibiotics.
* Mouth rinses other than the study drug.

Concurrent Treatment:

Excluded:

* Dental prophylaxis.

Patients with the following are excluded:

* Complete dentures, full partial dentures, removable dentures which fit poorly, or any prosthetic appliances which cannot be cleaned with sodium hypochlorite.
* Allergies to chlorhexidine.
* Sensitivity/intolerance to alcohol.
* Anterior composite/acrylic restorations with poor marginal adaption.
* Gross periodontal neglect or periodontal treatment within the past two weeks.
* Inability to comply with the study protocol based on the investigator's discretion.

Prior Medication:

Excluded within 7 days of study entry:

* Systemic or oral topical mucocutaneous antifungal therapy.
* Antibiotics.
* Daily use of mouth rinses.
* Excluded within 1 month of study entry:
* Systemic or oral topical corticosteroids.

Prior Treatment:

Excluded within 2 weeks of starting study drug:

* Dental prophylaxis or periodontal treatment.

Patients must be:

* HIV positive.
* Previously experienced at least one episode of clinically diagnosed oral candidiasis but currently free of clinical signs of oral candidiasis.
* Willing to sign informed consent.
* Willing to complete a medical history.

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Dental Research Institute / UCLA Med Ctr, Los Angeles, California
  - UCSF / Stomatology Clinical Ctr, San Francisco, California
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Bering Dental Clinic, Houston, Texas
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas

REFERENCES:
- [Background] Greenspan D. Treatment of oral candidiasis in HIV infection. Oral Surg Oral Med Oral Pathol. 1994 Aug;78(2):211-5. doi: 10.1016/0030-4220(94)90149-x. PMID 7936591